CLINICAL TRIAL: NCT02715414
Title: Family Groups for Urban Youth With Disruptive Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Silver School of Social Work (Other)
Responsible Party: Principal Investigator, Mary M. McKay, McSilver Professor of Poverty Studies, Director, McSilver Institute for Poverty Policy and Research, NYU Silver School of Social Work
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH106771 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-22 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Multiple Family Group (MFG) (Active Comparator): A multiple family group (MFG) is a 12-week, family-centered, group delivered intervention consists of six to eight families (caregiver/child dyads). Groups meet for approximately two hours per week, and sessions focus on targeting family-level factors that are associated with child problem behaviors. Specifically, eight of the 12 sessions are devoted to establishing rules (family organization, consistent discipline), responsibilities (inter-connectedness, expectancies), relationships (family warmth, within family support), respectful communication (family communication and conflict). An additional four sessions are focused on factors that impact the ability of families to incorporate new behaviors (family stress and social support).
  Interventions: Behavioral: MFG
- MFG + Clinic Implementation Team (Experimental): This condition consists of service providers, directors, and clinic staff who will create site-specific plans to enhance uptake and implementation of MFG. CITs address potential barriers to implementation and adjust the format and structure of MFG as needed in order to be implemented as part of clinic care.
  Interventions: Behavioral: Multiple Family Group + Clinic Implementation Team
- Standard Care (No Intervention): Standard Care consists of services including outpatient individual and family therapy, which are offered as part of clinic care.

INTERVENTIONS:
Behavioral: Multiple Family Group + Clinic Implementation Team — Clinic Implementation Teams (CIT) include providers at the clinic that aim to enhance uptake and implementation of MFG through modifications of MFG (e.g., format, length of sessions), but no modification to content will occur.
  Arms: MFG + Clinic Implementation Team
Behavioral: MFG — MFG is a 12-week group involving 6-8 families of children with problem behaviors. MFG aims to reduce family-level factors that are associated with the onset and perpetuation of problem behaviors. Eight of the 12 sessions are devoted to rules, responsibilities, respectful communication and relationships. Four additional sessions target family stress and social support.
  Other Names: Multiple Family Group
  Arms: Multiple Family Group (MFG)

SUMMARY:
A multiple family group (MFG) is a family-centered, group delivered, evidence-informed, manualized intervention that targets the most common reason for referral to publicly funded clinics: youth oppositional defiant and conduct disorders. This study will employ a mixed methods Type II effectiveness-implementation hybrid research design.In collaboration with the New York State Office of Mental Health (OMH), this longitudinal study will be conducted across the New York City (NYC) OMH licensed child behavioral health clinic system (n=134). The investigators will use mixed methods, and involve 268 providers and 2,688 adult caregivers of youth (7 to 11 years).

The following Specific Aims guide this study: To examine 1) short-term and longitudinal impact of MFGs on urban youth with Oppositional Defiant Disorder (ODD) and Conduct Disorder (CD) (replication); 2) family-level mediators (e.g. parenting, family process) of child outcomes; 3) clinic (readiness to adopt an innovation, leadership support and climate) and provider level moderators (preparedness, motivation and fidelity) of MFG implementation and integration and; 4) the impact of Clinic Implementation Teams (CIT) on clinic and provider level moderators of MFG implementation and integration. In this Randomized Controlled Trial, clinics will be stratified by borough (Manhattan, Queens, Bronx, Brooklyn, Staten Island) and randomly assigned within borough to 3 study conditions: 1) MFG+CITs; 2) MFG (with standard research training and consultation) or; 3) Standard Care. Data will be collected baseline, 8 and 16 weeks and 6 mo. follow-up) in Phase 1 (focus on implementation) and Phase II (integration).

DETAILED DESCRIPTION:
This study aims to generate knowledge needed to address seemingly intractable urban service delivery challenges: 1) lack of engagement of low-income youth with serious disruptive behavioral disorders and their families; 2) too few clinics offering family-based, evidence-informed services; 3) lack of scalable, empirically supported interventions designed for resource-strapped child settings and; 4) few empirically supported options for public policy makers to support the uptake and integration of service innovations in their systems.

A multiple family group (MFG) is a family-centered, group delivered, evidence-informed, manualized intervention that targets the most common reason for referral to publicly funded clinics: youth oppositional defiant and conduct disorders.5,6 MFGs target family factors which have been consistently implicated in the onset and maintenance of childhood behavioral disorders.7-9 and integrate components of existing evidence-based practices (EBPs). The MFG service delivery model was developed in collaboration with urban parents and service providers to address the serious challenges associated with EBP roll-outs: low rates of family involvement; poor uptake by providers; clinic and provider impediments to maintaining fidelity; and attenuated child outcome effects. These obstacles are pervasively associated with living and providing care within poverty-impacted communities and resource scarce, urban child behavioral health systems.

Findings from a recently completed NIMH-funded R01 trial, "Family Groups for Urban Youth with Disruptive Behavior" reveal that MFGs are associated with significant improvements relative to standard care (SC) in: 1) rates of family engagement and retention (80% completed); 2) short- (16 weeks) and long-term (10 months) improvements in child conduct problems and impairment; and 3) improvements in parenting and family processes. Although promising, this earlier study did not systematically examine specific mechanisms of family-level change hypothesized to influence child behavior.

Further, although the clinic directors (n=13) and MFG providers (n= 62) expressed strong endorsement of MFGs for their urban, resource constrained sites, significant implementation challenges emerged, potentially compromising future fidelity and sustainability. Thus, clinic and provider-level moderators of MFG implementation and integration will be examined in the current study. The proposed study will also examine a specific implementation strategy based on social-organizational theory (PRISM). Specifically, the investigators will experimentally test the impact of local child mental health clinic implementation teams (CITs), consisting of supervisors, service providers and family partners, on the implementation and integration of MFG. CITs will create site-specific plans to enhance multi-level implementation processes (e.g. clinic readiness to adopt an innovation, leadership support, provider preparedness, motivation and fidelity) in order to increase the likelihood of integrating MFGs into urban child behavioral health clinics.

The proposed study, in response to RFA 15-320, Clinical Trials to Test the Effectiveness of Treatment, Preventative, and Services Interventions, will employ a mixed methods Type II effectiveness-implementation hybrid research design. In collaboration with the NYS Office of Mental Health (OMH), this longitudinal study will be conducted across the NYC OMH licensed child behavioral health clinic system (n=134). The investigators will use mixed methods, and involve 268 providers and 2,688 adult caregivers of youth (7 to 11 years).

This study will examine:

1. short-term and longitudinal impact of MFGs on urban youth with ODD and CD (replication);
2. family-level mediators (e.g. parenting, family process) of child outcomes;
3. clinic (readiness to adopt an innovation, leadership support and climate) and provider level moderators (preparedness, motivation and fidelity) of MFG implementation (Phase I) and integration (Phase II);
4. the impact of CITs on clinic and provider level moderators of MFG implementation (Phase I) and integration (Phase II).

In this RCT, clinics will be stratified by borough (Manhattan, Queens, Bronx, Brooklyn, Staten Island) and randomly assigned within borough to 3 study conditions: 1) MFG+CITs; 2) MFG (with standard research training and consultation) or; 3) Standard Care. Data will be collected baseline, 8 and 16 weeks and 6 mo. follow-up) in Phase 1 (focus on implementation) and Phase II (integration).

The investigators team includes the highest level of NYSOMH research and policy leadership. McKay and Hoagwood are the co-Directors of the NYS Clinic Technical Assistance Center, the NIMH-funded Advanced Center on Implementation of Evidence-based Practice for Children in State Systems (IDEAS; P30 MH09032) and the Center for Collaborative Urban Child Mental Health Services Research (CCCR; P20 MH085983). Advanced methodological expertise (Jaccard, Palinkas), policy (Hogan, Bradbury, Goldman), family (Kuppinger) and provider (Cleek, Perri) consultation from IDEAS/CCCR Center advisors positions the study for maximum public health impact. This team is uniquely prepared to build on an existing research and service infrastructure within a state public mental health system to conduct this study. Because of the nationally-focused centers and the partnerships with NYSOMH, the findings from this study are immediately actionable.

ELIGIBILITY:
Inclusion criteria:

* provider willing to participate
* an adult caregiver of a child between 7 and 11 years of age with a diagnosis of Oppositional Defiant Disorder or Conduct Disorder

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2956 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Child Behavior and Impairment | Baseline, treatment mid-point (8 weeks), posttest (16 weeks), and six month followup (post-treatment)
  Child behavior and impairment is assessed via the Disruptive Behavior Disorders Rating Scale.

OTHER OUTCOMES:
Change in Family processes (e.g., rules, responsibilities, relationships, respectful communication) | Three times points: Baseline, treatment mid-point (8 weeks), posttest (16 weeks)
  Family processes, as measured by the Family Assessment Measure, are proposed to mediate primary outcomes
Change in Parent stress | Three times points: Baseline, treatment mid-point (8 weeks), posttest (16 weeks)
  Parent Stress, as measured by the Parenting Stress Index, are proposed to mediate primary outcomes
Change in Clinic readiness and leadership | Baseline and posttest (16 weeks)
  Measured via the Organizational Readiness for Change
Change in Clinic Climate | Baseline and posttest (16 weeks)
  Measured via the Community-Oriented Programs Environment Scale
Implementation of the intervention | Three times points: Baseline, treatment mid-point (8 weeks), posttest (16 weeks)
  Program Sustainability Assessment Tool
Change in Provider Motivation and Preparedness | Three times points: Baseline, treatment mid-point (8 weeks), posttest (16 weeks)
  MACS Process Measure.
Change in Child Behavior (assessed by Iowa Conners Rating Scale) | Four time points: baseline, treatment mid-point (8 weeks), posttest (16 weeks), and six month followup (post-treatment)
  Iowa Conners Rating Scale.
Change in Functional Impairment: Child (assessed by Impairment Rating Scale) | Four time points: baseline, treatment mid-point (8 weeks), posttest (16 weeks), and six month followup (post-treatment)
  Impairment Rating Scale
Fidelity to the intervention | Three times points: Baseline, treatment mid-point (8 weeks), posttest (16 weeks)
  Measured via the MFG Intervention Fidelity Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- McSilver Institute for Poverty Policy and Research - New York University Silver School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected in this project will be made available to the scientific community for educational, research, and non-profit purposes, and will meet the standards established by NIH and rigorous human subjects protection. Investigators in this proposal will adhere to NIH policy on data sharing as described in http://grants2.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm. Data request forms and procedures and policies for data sharing have been developed following these guidelines.

REFERENCES:
- [Background] Acri, M., Gopalan, G., Chacko, A., & McKay, M. (in press). Engaging families into treatment for child behavior disorders: A synthesis of the literature. In J. Lochman & W. Mathys (Eds.), Wiley Handbook of Disruptive and Impulse-Control Disorders.
- [Background] Hamovitch E, Acri M, Bornheimer LA. Who is accessing family mental health programs? Demographic differences before and after system reform. Child Youth Serv Rev. 2018 Jan;85:239-244. doi: 10.1016/j.childyouth.2017.12.027. Epub 2017 Dec 24. PMID 29736093
- [Background] Bornheimer, L. A., Acri, M., Parchment, T. ( in press). Attitudes towards and use of Evidence-Based Practice among providers of child mental health services in New York City. Research on Social Work Practice.
- [Result] Acri MC, Bornheimer LA, Jessell L, Chomancuzuk AH, Adler JG, Gopalan G, McKay MM. The intersection of extreme poverty and familial mental health in the United States. Soc Work Ment Health. 2017;15(6):677-689. doi: 10.1080/15332985.2017.1319893. Epub 2017 Jun 29. PMID 29618956
- [Derived] Acri M, Hamovitch E, Mini M, Garay E, Connolly C, McKay M. Testing the 4Rs and 2Ss Multiple Family Group intervention: study protocol for a randomized controlled trial. Trials. 2017 Dec 4;18(1):588. doi: 10.1186/s13063-017-2331-7. PMID 29202867